CLINICAL TRIAL: NCT04377191
Title: Comparison of The Effect of Two Different Virtual Reality Trainings on Gait, Balance and Posture of Individuals With Dementia
Brief Title: The Effect of Different Virtual Reality Trainings on Gait, Balance and Posture of Individuals With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-65; 5444 (Other Grant/Funding Number: Ankara Yildirim Beyazit University Scientific Research Projects Office)
Record Dates: First submitted 2020-05-02; First posted 2020-05-06 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Dementia
Keywords: dementia; virtual reality; exergame; gait
MeSH Terms: conditions — Dementia | interventions — Exergaming; Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VR 1 Group (Experimental): In this group, participants received standard exercise and exergame training with Microsoft Xbox 360 Kinect for 2 days per week for 6 weeks.
  Interventions: Other: exergame; Other: exercise
- VR 2 Group (Experimental): In this group, participants received standard exercise and exergame training with ALDA balance gear for 2 days per week for 6 weeks.
  Interventions: Other: exergame; Other: exercise
- Control Group (Active Comparator): In this group, participants received only standard exercise for 2 days per week for 6 weeks.
  Interventions: Other: exercise

INTERVENTIONS:
Other: exergame — Microsoft Xbox 360 Kinect The exercises were advanced from simple to complex. The program started with exercises in a sitting position. In the next stage, the games requiring weight transfer and use of upper limbs in standing position were continued. The program ended with games that require more complex movements such as lunge and mini squats.
  Other Names: virtual reality; Microsoft Xbox 360 Kinect
  Arms: VR 1 Group
Other: exergame — ALDA In the training, games that could be controlled by balance swing, trunk movements and weight transfer in sitting or standing position were used.
  Other Names: virtual reality; ALDA
  Arms: VR 2 Group
Other: exercise — Standard Exercise Program The program included warm-up, main exercise and cooling. Warm-up and cooling included neck, trunk, upper-lower extremity range of movement (ROM) exercises and stretching exercises. Main exercise included postural alignment, strengthening for trunk and lower extremity, balance and walking exercises.

SUMMARY:
Dementia, a part of geriatric syndrome, is characterized by the deterioration of multiple cognitive domains such as memory, language, orientation, learning and personality as a result of damage to the central nervous system and in terms prognosis persistent and often progressive clinical condition. In the epidemiological studies it is stated that the number of the dementia affected people approximately 2 times in every 20 years. In several studies, it has been mentioned that cognitive disorders affect individuals' motor function such as gait and postural responses. These effects lead to a vicious circle by causing immobilization of individuals due to a decrease in cognitive functions in addition to immobilization due to aging. The lack of pharmacological therapies to change the prognosis of dementia, emphasizes physical activity methods due to its neurological contributions. However, due to the fact that conventional exercise programs are seen as boring in terms of elderly individuals and the exercise attendance rates are low, the virtual reality (VR) training have been preferred recently. To the best of the investigator's knowledge, there is no study examining the effect of different virtual reality trainings on the spatio-temporal characteristics of the gait, posture and balance. Therefore, the aim of this study is to evaluate the effect of different virtual reality trainings on these parameters.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with dementia
* Mini-Mental State Examination (MMSE) score between 18-23 points
* Able to walk independently with/without a walking aid (a single point cane)
* Able to speak and understand Turkish
* Understand simple commands
* At least primary education

Exclusion Criteria:

* Severly vision and hearing problems
* Undergo acute retinal hemorrhage or ophthalmic surgery
* Acute or chronic neurological problems
* Musculoskeletal and/or neurological problems affecting movement and balance
* Vestibular problem and/or use medicine
* Uncontrolled cardiovascular disease, congestive heart failure, acute myocarditis, pulmonary hypertension, or using a pacemaker
* Malignancy
* Orthopedic or neurological surgery in the past 6 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-11-09 (Actual); Study Completion 2019-12-24 (Actual)

PRIMARY OUTCOMES:
gait speed | change from baseline at 6 weeks
  Gait speed was assessed by BTS G-Walk inertial sensor. The sensor, connected to the Lumbal 4-5 intervertebral space via a semi-elastic belt, transfers the spatiotemporal characteristics of the gait to the computer via Bluetooth® 3.0 (G-Studio® software). In our study, participants were asked to walk in a corridor of 8 meters.

SECONDARY OUTCOMES:
Spatiotemporal Characteristics of Gait | change from baseline at 6 weeks
  Spatiotemporal characteristics of gait was assessed by BTS G-Walk inertial sensor. The assessed characteristics were cadence, stride length, left and right step length, step length/height ratio, gait cycle time,stance phase %, swing phase%, double support %, single support %. The sensor, connected to the Lumbal 4-5 intervertebral space via a semi-elastic belt, transfers the spatiotemporal characteristics of the gait to the computer via Bluetooth® 3.0 (G-Studio® software). In our study, participants were asked to walk in a corridor of 8 meters.
Berg Balance Scale | change from baseline at 6 weeks
  Berg Balance Scale (BBS) was used to evaluate static balance ability.It is a widely used and validated scale for elderly people. Validity and reliability of BBS in Turkish was established by Sahin et al. The scale includes 14 functional activities such as transfers, turning, taking objects from the ground. Each activity scores between 0-4 and high scores indicate good balance ability.
Timed Up and Go Test | change from baseline at 6 weeks
  Timed Up and Go Test (TUGT) was used to assessed dynamic balance ability. Participants were asked to stand up from the chair, walk 3 meters and go back and sit on the chair. Performance time recorded in seconds.
New York Posture Scale | change from baseline at 6 weeks
  New York Posture Scale was used to evaluate upright posture. It evaluates head, shoulders, spine, hip and foot alignment in the frontal plane. It evaluates head, thorax, shoulders, upper thoracic region, trunk, abdomen and lower lumbar region alignment in the sagittal plane. In total, 13 regions are evaluated. Each item on the scale gets 1, 3 or 5 points depending on the degree of deviation from the normal. High scores represent a good posture.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)